CLINICAL TRIAL: NCT06637748
Title: Echo and Electrocardiographic Findings in Children With Bronchial Asthma At Sohag University Hospital
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Safa Atef Abodaif, Resident-pediatric department-sohag hospital university, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: soh-Med-24 - 09- 04MS
Record Dates: First submitted 2024-10-08; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Bronchial Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acute Exacerbation Group (Active Comparator): an acute attack, at least 1 month after attack. a. Mild acute exacerbation b. Moderate acute exacerbation c. Severe acute exacerbation, according GINA 2024.
  Interventions: Procedure: Echocardiography; Procedure: Electrocardiography
- Stable Asthma Group (Active Comparator): Patients attending routine follow-up visits with well-controlled asthma
  Interventions: Procedure: Echocardiography; Procedure: Electrocardiography

INTERVENTIONS:
Procedure: Echocardiography — Transthoracic echocardiography
  • Parameters assessed:
  * Right ventricular dimensions and function
  * Pulmonary artery pressure estimation
  * Valvular function assessment
  * Left ventricular dimensions (end-diastolic and end-systolic)o Left ventricular function (ejection fraction, fractional shortening)
Procedure: Electrocardiography — Standard 12-lead ECG recording
  • Parameters assessed:
  * Heart rate and rhythm
  * P-wave morphology
  * PR interval
  * QRS complex duration and morphology
  * ST-segment changes
  * T-wave abnormalities
  * QT interval

SUMMARY:
Bronchial asthma is a common respiratory disorder among children, worldwide. Asthma is characterized by chronic inflammation and remodeling of the airways induced by recurrent exposure to hypoxemia that leads to repeated tissue injury and repair. The interaction between respiratory diseases and cardiovascular function is complex . Cardiac dysfunction can be attributed to pulmonary hypertension (PH) secondary to recurrent hypoxia in patients with bronchial asthma. PH affects the pulmonary vasculature by releasing various cytokines leading to pulmonary vasoconstriction and enhancing the remodeling process with muscularization and proliferation of the vascular media and intima . Other hypotheses concluded that the exaggerated respiratory efforts may raise the intrathoracic pressure and increase right ventricle (RV) afterload and consequently RV hypertrophy and/or dilatation . Children with severe bronchial asthma can experience cor pulmonale later in life, but little is known about the early cardiac changes that might be present during childhood especially for mild or moderate persistent asthma. Some studies have reported right ventricular dysfunction as the earliest hemodynamic change among those cases . Other studies did not report these results and reported impaired systolic function of the left ventricle (LV) even before diastolic dysfunction . Insufficient control of BA, in turn, can cause the formation of various pathological conditions. For example, there are studies showing the risk of cardiac arrhythmias and conduction disorders in patients with uncontrolled BA due to functional changes or pathological remodeling of the myocardium . Atrial remodeling, which is the pathomorphological basis of serious supraventricular cardiac arrhythmias, has a more rapid progression with poor BA control and is formed as a result of excessive stretching of the atrial wall, as well as other adverse factors . The connection between BA and supraventricular arrhythmias, including atrial fibrillation (AF), was noted in studies by Cepelis et al. Available data indicate that in the adult population, cardiac arrhythmias are significantly more common in patients with BA than in those without it (9). The results of a Norwegian population study HUNT study, demonstrate that the risks of supraventricular arrhythmias and AF are increased in patients with an uncontrolled BA . Electrocardiography (ECG) is the universal screening method for assessing the state of the atrial myocardium and the conducting system of the heart. According to German et al. ECG analysis can make a significant input to the assessment of the risk of formation of supraventricular rhythm and conduction disorders. Therefore, the analysis of the atrial component of the ECG, and atrioventricular conduction in patients with BA is an important component of the management of these patients, especially in pediatric practice. Consequently, the study of the characteristics of the ECG and its supraventricular component in children with BA is relevan

ELIGIBILITY:
Inclusion Criteria:

* 1. Age range: 5-18 years 2. Confirmed diagnosis of bronchial asthma, made in accordance with current international and national consensus documents

Exclusion Criteria:

* . Known congenital heart disease 2. Presence of acute infectious diseases and fever 3. Diabetes 4. Autoimmune disorders 5. Primary immunodeficiency 6. Cancer 7. Current use of oral glucocorticoids 8. Other chronic respiratory conditions 9. Systemic diseases affecting the cardiovascular system

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Changes in ECG parameters from baseline to follow-up | 1 year
  Standard 12-lead ECG recording
  • Parameters assessed:
  * Heart rate and rhythm
  * P-wave morphology
  * PR interval
  * QRS complex duration and morphology
  * ST-segment changes
  * T-wave abnormalities
  * QT interval

SECONDARY OUTCOMES:
Changes in echocardiographic parameters from baseline to follow-up | 1year
  Transthoracic echocardiography
  • Parameters assessed:
  * Right ventricular dimensions and function
  * Pulmonary artery pressure estimation
  * Valvular function assessment
  * Left ventricular dimensions (end-diastolic and end-systolic)
  * Left ventricular function (ejection fraction, fractional shortening)

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

REFERENCES:
- [Background] Harkness LM, Kanabar V, Sharma HS, Westergren-Thorsson G, Larsson-Callerfelt AK. Pulmonary vascular changes in asthma and COPD. Pulm Pharmacol Ther. 2014 Dec;29(2):144-55. doi: 10.1016/j.pupt.2014.09.003. Epub 2014 Oct 12. PMID 25316209
- [Background] Wang X, Liu C, Wu L, Zhu S. Potent ameliorating effect of Hypoxia-inducible factor 1alpha (HIF-1alpha) antagonist YC-1 on combined allergic rhinitis and asthma syndrome (CARAS) in Rats. Eur J Pharmacol. 2016 Oct 5;788:343-350. doi: 10.1016/j.ejphar.2016.07.040. Epub 2016 Aug 4. PMID 27498367
- [Background] German DM, Kabir MM, Dewland TA, Henrikson CA, Tereshchenko LG. Atrial Fibrillation Predictors: Importance of the Electrocardiogram. Ann Noninvasive Electrocardiol. 2016 Jan;21(1):20-9. doi: 10.1111/anec.12321. Epub 2015 Nov 2. PMID 26523405
- [Background] Gordina AV, Egoshina KA, Eliseeva TI, Vinogradova NG, Ovsyannikov DY, Tush EV, Prakhov AV, Daniel-Abu MI, Khaletskaya OV, Kubysheva NI. The Relationship Between Bronchial Patency and Parameters of ECG Supraventricular Component in Children With Bronchial Asthma. Front Pediatr. 2020 Sep 16;8:576. doi: 10.3389/fped.2020.00576. eCollection 2020. PMID 33042919